CLINICAL TRIAL: NCT04014426
Title: Evaluation of Oxaliplatin Exposure and Security of Healthcare Workers During Pressurized Intraperitoneal Aerosol Chemotherapy
Brief Title: Evaluation of Healthcare Workers Safety During Pressurized Intraperitoneal Aerosol Chemotherapy
Acronym: PIPAC-Secure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC 2017/36
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Safety; Healthy Volunteers
Keywords: Peritoneal Carcinomatosis; Healthcare Workers; Security; Pressurized Intraperitoneal Aerosol Chemotherapy; Aerosols/administration & dosage; Oxaliplatin
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Exposed/ Non-exposed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed (Other): Healthcare workers participating at two PIPAC
  Interventions: Other: Blood sample; Other: Urinary sample
- Non-exposed (Other): Healthy volunteers unexposed to chemotherapy
  Interventions: Other: Blood sample; Other: Urinary sample

INTERVENTIONS:
Other: Blood sample — Exposed group:
  * 15 to 30 minutes before the start of the procedure: 1 EDTA tube of 6 ml for blood (T0)
  * 2hours after the end of the procedure: 1 EDTA tube of 6 ml (T1)
  Non-exposed group:
  - During the morning (8 to 10 a.m): 1 EDTA tube of 6 ml (T0)
Other: Urinary sample — Exposed group:
  * 15 to 30 min before the PIPAC procedure (T0)
  * 2hours after the end of the procedure (T1)
  * The next morning after the procedure (T2)
  Non-exposed group:
  - During the morning (8 to 10 a.m) (T0)

SUMMARY:
Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a new treatment that applies chemotherapeutic drugs into the peritoneal cavity as an aerosol. It is used to treat patient with Peritoneal Carcinomatosis (PC). During this procedure, healthcare workers may be under risks of exposure to cytotoxic treatments.

The purpose of this study is to evaluate the safety of the heathcare workers and the risk of operation room Oxaliplatin's contamination during a PIPAC.

DETAILED DESCRIPTION:
Peritoneal carcinomatosis (PC), which was long considered as a terminal stage, is now potentially curable. Nevertheless, in most cases, the surgical treatment of PC is limited by the disease extent which is commonly measured with the Peritoneal Carcinomatosis Index (PCI). For the patients that are not considered good candidates for resection, there are very few alternatives. Systemic chemotherapy may have limited or no effect therefore an alternative solution is needed for these patients.

Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a new treatment that applies chemotherapeutic drugs into the peritoneal cavity as an aerosol under pressure through minimal laparoscopic surgery.

Nevertheless, as it is the case for most technologies, security is not always completely tested. The innovative team started by establishing a set of security rules that concern the operating room ventilation, distance monitoring of the patient during nebulization, evacuation of the aerosols in a closed system. In a work dedicated to occupational hazards, the authors followed the following steps: identification of hazardous substances and dose; identification of possible exposure ways; simulation of the PIPAC procedure with nontoxic aerosols and smoke; redaction of standard operating procedures (SOP); second simulation according to the SOP; informing and training the health care workers; and performance of the first two PIPAC procedures with chemotherapeutic substances and workplace measurements under real conditions. At the end of the study, there were no traces of doxorubicin or cisplatin (the two drugs used in the two consecutive test procedures) in the operating room air, neither to the position of the anesthesiologist, nor of the surgeon.

This study does not concern PIPAC with oxaliplatin, nor does it research the presence of the drugs in the health caregivers.

Therefore we considered mandatory to further investigate occupational hazards in the specific case of oxaliplatin by focusing more on the healthcare workers and partially applying the same protocols as in the case of Heated intraperitoneal chemotherapy (HIPEC).

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects ≥ 18 and ≤ 70 years old

* Exposed subjects: The healthcarers involved in two different PIPAC using oxaliplatin (Surgeon, Anesthesiste, Block nurse …)
* Non-exposed subjects: Healthy volunteers not exposed to oxaliplatin or other platin based chemotherapy (administrative function).
* Must be affiliated to a social security system
* Informed consent agreement and signature

Exclusion Criteria:

* Legal incapacity or physical, psychological or mental status interfering with the subject's ability to sign the inform consent or to terminate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Blood levels of oxaliplatin - Exposed group | Change from before PIPAC and 2hours after PIPAC
  Blood levels of oxaliplatin in healthcare workers in two PIPAC
Blood levels of oxaliplatin - Non-exposed group | At baseline
  Blood levels of oxaliplatin in heathy subject non-exposed to chemotherapy
Urinary levels of oxaliplatin - Exposed group | Change from before PIPAC, 2hours after PIPAC and the next day after PIPAC
  Urinary levels of oxaliplatin in healthcare workers in two PIPAC
Urinary levels of oxaliplatin - Non-exposed group | At baseline
  Urinary levels of oxaliplatin in heathy subject non-exposed to chemotherapy

SECONDARY OUTCOMES:
Oxaliplatin contamination of the operating room | Before PIPAC and 10min after PIPAC
  Oxaliplatin dosed on standardized gazes used to clear four different spots in the operating room: the ceiling lamp, the electroagulation device, the laparoscopy tower and the anesthesia monitoring screen

CONTACTS AND LOCATIONS:
Overall Officials: Olivia SGARBURA, MD, Study Chair — ICM - Institut régional du Cancer Montpellier
Locations (1):
- ICM - Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tempfer CB, Celik I, Solass W, Buerkle B, Pabst UG, Zieren J, Strumberg D, Reymond MA. Activity of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin and doxorubicin in women with recurrent, platinum-resistant ovarian cancer: preliminary clinical experience. Gynecol Oncol. 2014 Feb;132(2):307-11. doi: 10.1016/j.ygyno.2013.11.022. Epub 2013 Nov 23. PMID 24275155
- [Background] Markman M. Intraperitoneal antineoplastic drug delivery: rationale and results. Lancet Oncol. 2003 May;4(5):277-83. doi: 10.1016/s1470-2045(03)01074-x. PMID 12732164
- [Background] Solass W, Giger-Pabst U, Zieren J, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy (PIPAC): occupational health and safety aspects. Ann Surg Oncol. 2013 Oct;20(11):3504-11. doi: 10.1245/s10434-013-3039-x. Epub 2013 Jun 14. PMID 23765417
- [Derived] Larroque M, Arnaudguilhem C, Bouyssiere B, Quenet F, Bouazza N, Jarlier M, Boulabas S, Mounicou S, Sgarbura O. Evaluation of the environmental contamination and exposure risk in medical/non-medical staff after oxaliplatin-based pressurized intraperitoneal aerosol chemotherapy. Toxicol Appl Pharmacol. 2021 Oct 15;429:115694. doi: 10.1016/j.taap.2021.115694. Epub 2021 Aug 21. PMID 34428445